CLINICAL TRIAL: NCT01977664
Title: The Factors Primarily Intrinsic to the Oocyte Are Responsible to the Oocyte Maturation Defective: a Case Report.
Brief Title: In Vitro Maturation Induction of Oocytes From a Woman With Syndrome of Repeated Oocyte Maturation Failure in Vitro
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yang Jie, Principal Investigator, The Second Affiliated Hospital of Kunming Medical University
Other Study IDs: 201301
Record Dates: First submitted 2013-10-09; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Oocyte Maturation Failure
Keywords: oocyte maturation failure; Maturation induction in vitro

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- oocyte maturation failure: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Donated oocytes is from a patient with repeated oocyte maturation failure in IVF cycles. Cytoplasm of matured metaphase II oocyte and active MPF were injected into the donated oocytes.

DETAILED DESCRIPTION:
The study reported a woman with syndrome of repeated oocyte maturation failure where there is repeated production of immature oocytes.She underwent two IVF cycles in other hospital. All oocytes obtained were immature and the treatment were stopped.She underwent her third try in our hospital. The couple gave their informed consent: ICSI will be performed if maturation occurred, otherwise, the treatment would be stopped and the oocytes would be donated for study if the oocytes were not matured after 24 hours of culture. After ovarian hyperstimulation,14 oocytes were obtained. None of them was matured. The cycle was canceled and the oocytes were donated for study.To induce the immature oocytes in vitro, oocytes were 1)cultured in follicular fluid containing matured metaphase II oocyte; 2) performed intracytoplasmic sperm injection (ICSI) to induce intracellular Ca2+]i oscillations; 3)injected with active maturation promoting factor (MPF), 4)injected with cytoplasm of matured metaphase II oocyte.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of syndrome of repeated oocyte maturation

Exclusion Criteria:

patients with matured oocytes in IVF cycles

Ages: 32 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: a patient with repeated oocyte maturation failure in IVF cycles
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Oocyte nucleus maturation | April，2012

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, M.Sc, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China